CLINICAL TRIAL: NCT00298896
Title: Phase 2 Open-Label, Multicenter Clinical Study of the Safety and Efficacy of Intravenous Administration of SNS-595 in Patients With Advanced Small Cell Lung Cancer (SCLC)
Brief Title: Safety and Efficacy Clinical Study of SNS-595 in Patients With Advanced Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0006
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma, Small Cell; Small Cell Lung Cancer
Keywords: Lung; Squamous Cell; Small Cell; Carcinoma; Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma; Carcinoma; Neoplasms | interventions — vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNS-595 (Experimental): SNS-595; 48 mg/m2 administered IV once every 21 days for up to 6 cycles.
  Interventions: Drug: SNS-595

INTERVENTIONS:
Drug: SNS-595
  Other Names: Voreloxin; Vosaroxin

SUMMARY:
The purpose of this study is to evaluate the objective tumor response rate to SNS-595 in patients with small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
Other objectives of this study are to assess the safety, survival rate, best response, time to disease progression, duration of tumor response, and to explore several potential biomarkers to see how these levels change after administration of SNS-595.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign a written informed consent document
* Patients who have recurrent or refractory SCLC requiring second-line chemotherapy who previously received first-line chemotherapy
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Brain metastasis may be included if the patient is neurologically stable and has been off steroids and anticonvulsants for at least 4 weeks prior to Cycle 1 Day 0
* Laboratory values within the normal or reasonable reference range as specified by the protocol

Exclusion Criteria:

* Prior exposure to SNS-595
* Pregnant or breastfeeding
* Women of childbearing potential, or male partners of women of childbearing potential, unwilling to use an approved, effective means of contraception according to the institution's standards
* Other active malignancies or other malignancies within the past 12 months, other than non-melanoma skin cancer, cervical intraepithelial neoplasia, or prostatic intraepithelial neoplasia
* Q-wave myocardial infarction or cerebrovascular accident/transient ischemic attack (TIA) within 6 months before the first SNS-595 dose
* Thromboembolic event (deep vein thrombosis or pulmonary embolus) within 28 days before the first SNS-595 dose
* Requires kidney dialysis (hemodialysis or peritoneal)
* Prior chemotherapy, investigational agents, or radiation therapy within 28 days before Cycle 1 Day 0; however, nitrosoureas, mitomycin C, and therapeutic monoclonal antibodies are not permitted for at least 42 days before Cycle 1 Day 0
* In patients with toxicities caused by prior cancer therapy, those toxicities must have returned to less than or equal to Grade 1, with the exception of alopecia.
* Prior pelvic radiation therapy or radiation to greater than 25% of bone marrow reserve; radiation to the brain is permitted up to 28 days before the first SNS-595 dose, as long as the patient does not require treatment with corticosteroids for symptom control related to brain metastases.
* Any other medical, psychological, or social condition that, in the opinion of the Principal Investigator, would contraindicate the patient's participation in the clinical trial due to safety or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Berman, MD, Study Director — Sunesis Pharmaceuticals
Locations (17):
- United States (12):
  - University of California Davis, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Laval, Sainte-Foy, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNS-595
Started | 55
Completed | 5
Not Completed | 50
Not completed — Death | 3
Not completed — Physician Decision | 2
Not completed — Intercurrent Illness | 1
Not completed — Disease Progression | 41
Not completed — Withdrawal by Subject | 2
Not completed — Assigned to treatment in error | 1

BASELINE CHARACTERISTICS:
Population: Patients with advanced platinum-sensitive or refractory small cell lung cancer (SCLC) requiring second-lie chemotherapy after prior first-line therapy.
Arm/Group | SNS-595
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 54
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 14
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective tumor response rate based on the RECIST criteria for target lesions as assessed by CT or MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD), at least a 20% increase in the sum of the LD of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Overall Response (OR) = CR + PR
Time Frame: up to 6 months
Population: Efficacy Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | SNS-595
Number analyzed (Participants) | 47
Participants | 3

2. Secondary Outcome: Best Overall Response
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started), classified as CR, PR, SD or PD per RECIST criteria.
Time Frame: upto 6 months
Population: Efficacy Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | SNS-595
Number analyzed (Participants) | 47
Participants
  Complete Response | 1
  Partial Response | 2
  Progressive Disease | 31
  Stable Disease | 13

ADVERSE EVENTS:
Time Frame: From time of first dosing of study treatment (up to 6 cycles of 21 days each) to 28 days post last treatment, i.e., approximately 5.1 months.
Description: One enrolled patient removed from assessment due to error in admission to study (prior to study drug administration) and is therefore not included in the "Participants at Risk" data (54 of 55 participants).
Groups:
- SNS-595: SNS-595; 48 mg/m2 administered IV once every 21 days for up to 6 cycles.
  SNS-595
Arm/Group | SNS-595
All-Cause Mortality (participants affected / at risk) | 15/54
Serious Adverse Events (participants affected / at risk) | 9/54
Other Adverse Events (participants affected / at risk) | 52/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNS-595 (N=54)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sudden death (General disorders) | 1
Pneumonia (Infections and infestations) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNS-595 (N=54)
Anaemia (Blood and lymphatic system disorders) | 9
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 4
WBC abnormal (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blindness transient (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Breath odour (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 28
Odynophagia (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 9
Chest discomfort (General disorders) | 1
Chills (General disorders) | 4
Disease progression (General disorders) | 6
Fatigue (General disorders) | 39
Gait disturbances (General disorders) | 1
General physical health deterioration (General disorders) | 1
Hyperhidrosis (General disorders) | 2
Influenza like illness (General disorders) | 1
Lethargy (General disorders) | 1
Mucosal inflammation (General disorders) | 4
Nodule (General disorders) | 1
Non-cardiac chest pain (General disorders) | 8
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 4
Pitting oedema (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Blister (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Breath sounds abnormal (Investigations) | 1
Weight decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 10
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercalcaemia of malignancy (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5
Polydipsia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Akathisia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 8
Memory impairment (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Restlessness (Psychiatric disorders) | 1
Bladder distension (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Urine abnormality (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Plerual effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Further study is needed to confirm the results due to limited sampling size. Statistical fields are not included here because no statistical testings were performed to compare any of the treatment groups. No p-values or odds ratios were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days